CLINICAL TRIAL: NCT05436925
Title: Improving Growth and Neurodevelopmental Outcomes in Preterm Infants Experiencing Hyperglycemia
Brief Title: CGM Use in Preterm Infants
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2022-30647
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Very Low Birth Weight Infant; Very Preterm Maturity of Infant; Hyperglycemia
Keywords: Continuous glucose monitor; Neonates; Hyperglycemia; Hypoglycemia; Very low birth weight
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Dexcom G6 sensor Continuous Glucose Monitor (CGM): All participants will be assigned to use the continuous glucose monitor
  Interventions: Device: Dexcom G6 sensor Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Dexcom G6 sensor Continuous Glucose Monitor (CGM) — The device used as part of the study is to obtain results for glucose testing for research only and not for diagnostic purposes.

SUMMARY:
Preterm infants (gestational age (GA) at birth < 31 weeks) admitted to the University of Minnesota Masonic Children's Hospital NICU will have a Dexcom G6 sensor Continuous Glucose Monitor (CGM) placed shortly after consent and wear the device for up to 10 days. The low alarm threshold will be set at 60 mg/dL or 80mg/dL (depending on whether they are receiving continuous insulin) to detect the potential for hypoglycemia. A suggestion will be made to the clinical team to draw a blood glucose to correlate with CGM values ≤60 mg/dL and the infant will be treated according to Neonatal Intensive Care Unit (NICU) protocol for corroborating blood glucose levels. Infants will also be monitored per current NICU protocol (blood glucose checks every 1-2 hours while on insulin) and treated accordingly. Clinical data and long-term growth, body composition and neurodevelopmental outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants (gestational age (GA) at birth < 31 weeks)
* admitted to the University of Minnesota Masonic Children's Hospital Neonatal Intensive Care Unit
* written informed consent can be secured from a parent within 96 hours of birth.

Exclusion Criteria:

* Infants born at ≥31 weeks GA
* infants with a prenatally diagnosed clinical or genetic condition (other than prematurity) that is known to affect growth rate, adiposity, or neurocognitive development
* children experiencing severe birth asphyxia,
* children enrolled in another nutritional study,
* children likely to be transferred out of the NICU

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants (gestational age (GA) at birth <31 weeks) admitted to the University of Minnesota Masonic Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Detection of hypo- and hyperglycemia - CGM device | 10 days post placement of CGM
  Proportion of CGM device readings that match blood glucose readings
Detection of hypo- and hyperglycemia - 60 mg/dL | 10 days post placement of CGM
  % time below 60 mg/dL
Detection of hypo- and hyperglycemia - 180 mg/dL | 10 days post placement of CGM
  % time above 180 mg/dL
Detection of hypo- and hyperglycemia - AEs | 10 days post placement of CGM
  % of infants with adverse events secondary to CGM placement or wear

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States